CLINICAL TRIAL: NCT01110408
Title: A Prospective, Randomized, Double-Blind, Multicenter Study to Establish the Safety and Tolerability of Doripenem Compared With Cefepime in Hospitalized Children With Complicated Urinary Tract Infections
Brief Title: A Safety and Tolerability Study of Doripenem Compared With Cefepime in Children Hospitalized With Complicated Urinary Tract Infections
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Trial terminated early per business decision
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR016792; DORIPED3002 (Other: Janssen Research & Development, LLC); 2009-015953-18 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2010-04-15; First posted 2010-04-26 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Complicated Urinary Tract Infections or Pyelonephritis
Keywords: Antibiotic; Child, Hospitalized; Complicated Urinary Tract Infection; Pyelonephritis; Doripenem; Cefepime
MeSH Terms: conditions — Pyelonephritis | interventions — Doripenem; Cefepime; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doripenem (Experimental): Doripenem 20 mg/kg per dose (up to 500 mg/dose) will be administered every 8 hours as 60-minutes IV (at least 3 days of IV doripenem only or IV doripenem followed by oral amoxicillin/clavulanate potassium or ciprofloxacin). Total duration of treatment 10 to 14 days.
  Interventions: Drug: Doripenem; Drug: Cefepime placebo; Drug: Amoxicillin/clavulanate potassium
- Cefepime (Experimental): Cefepime 50 mg/kg per dose (up to 2 g/dose) will be dministered every 8 hours as 30-minutes IV (at least 3 days of IV cefepime only or IV cefepime followed by oral amoxicillin/clavulanate potassium or ciprofloxacin). Total duration of treatment 10 to 14 days.
  Interventions: Drug: Doripenem placebo; Drug: Cefepime; Drug: Amoxicillin/clavulanate potassium

INTERVENTIONS:
Drug: Doripenem — Type=once every 8 hours infused over 60 minutes, Unit=mg,Number=20mg/kg up to 500mg/dose, Form=solution for infusion,Route=intravenous use. At least 3 days of iv doripenem administered every 8 hours immediately after each iv infusion of cefepime placebo for up to 14 days
  Arms: Doripenem
Drug: Doripenem placebo — Form=solution for infusion, Route=intravenous use, administered once every 8 hours infused over 60 minutes immediately following each iv infusion of cefepime for up to 14 days
  Arms: Cefepime
Drug: Cefepime — Type=once every 8 hours, Unit=mg, Number=50 mg/kg up to 2g/dose, Form=solution for infusion, Route=intravenous use. At least 3 days of iv cefepime administered every 8 hours infused over 30 minutes immediately before each iv infusion of doripenem placebo for up to 14 days
  Arms: Cefepime
Drug: Cefepime placebo — Form=solution for infusion, Route=intravenous use, administered once every 8 hours infused over 30 minutes immediately before each iv infusion of doripenem for up to 14 days
  Arms: Doripenem
Drug: Amoxicillin/clavulanate potassium — Form=suspension or tablets, Route=oral (by mouth), may be administered at the discretion of the investigator once every 12 hours for up to 14 days following IV therapy with doripenem or cefepime.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of doripenem compared to cefepime in children hospitalized with complicated urinary tract infections.

DETAILED DESCRIPTION:
This is a randomized (study assigned by chance), double-blind (neither physician nor patient knows the name of the assigned study drugs), double-dummy (all patients are given both a placebo [salt solution] and study drug in alternating periods of time during the study), active comparator-controlled (compare the 'test' treatment to standard-of-care therapy), multinational, multicenter study to establish the safety and tolerability of the antibiotic doripenem compared with the antibiotic cefepime administered by intravenous (iv) infusion (slow injection of drug solution into the vein over a period of time) in children ages 3 months to less than 18 years hospitalized with a complicated urinary tract infection (cUTI). The study includes 3 periods: a pretreatment (screening) period that will occur within 2 days prior to randomization (assignment of study drug); a treatment period of 10 to 14 days where the patients will receive study drug treatment, and a posttreatment period consisting of 2 study visits. The maximum duration of study drug therapy is 14 days. The total duration of the study is approximately 7 to 8 weeks for each patient. Safety and tolerability will be evaluated by examining the incidence, severity, and type of adverse events, changes in clinical laboratory tests, vital sign measurements, and findings from physical examinations that are recorded as adverse events during treatment and at each posttreatment visit. An independent monitoring committee (IDMC) will be established for this study to ensure that the safety of patients is not compromised. The IDMC will consist of individuals who are not associated with the conduct of the study, and will include but will not be limited to individuals with expertise relevant to the care of pediatric patients, and including at least one infectious disease physician and at least one statistician. IV study drug therapy (Cefepime [50mg/kg up to 2g/dose] and doripenem placebo or doripenem [20mg/kg up to 500mg/dose] and cefepime placebo will be administered once every 8 hours for up to 14 days. After receiving a minimum of 3 days of IV study drug therapy, patients may be discharged from the hospital and continue PO antibiotic therapy with amoxicillin/clavulanate potassium, ciprofloxacin, or alternative antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are eligible for the study must have a current episode of cUTI or pyelonephritis
* Have evidence of pyuria that meets criteria specified in the study protocol
* Have a study-qualifying pretreatment "baseline" urine culture specimen obtained by an acceptable method within 48 hours before the start of the administration of the first dose of iv study drug from which a bacterial pathogen is isolated with a growth of >= 100000 colony forming units (CFU)/mL
* Require hospitalization initially and 10 to 14 days of antibacterial therapy [of which at least 72 hours should be iv therapy] for the treatment of the presumed UTI
* Have a signed informed consent form completed by the patient's parent or legal representative (and a signed assent form obtained from patients who are capable of providing assent, typically, children 7 years of age or older)

Exclusion Criteria:

* Have a history of hypersensitivity reactions to carbapenems, cephalosporins, penicillins, or other beta-lactam antibiotics
* concomitant infection including but not limited to suspected or confirmed meningitis or central nervous system infection requiring systemic antibiotic or antifungal therapy in addition to the iv study drug therapy at the time of randomization
* Receipt of any amount of systemic antibiotic within 96 hours before obtaining the study-qualifying pretreatment baseline urine or systemic antibiotic therapy for more than 24 hours after obtaining the study-qualifying pretreatment baseline urine specimen
* Have a diagnosis of intractable UTI/pyelonephritis infection anticipated to require more than 14 days of study drug therapy, a permanent indwelling bladder catheter or instrumentation including nephrostomy or current urinary catheter that will not be removed or anticipation of urinary catheter placement that will not be removed during the course of iv study drug therapy administration, complete and permanent obstruction of the urinary tract, confirmed fungal UTI, suspected or confirmed perinephric or intrarenal abscess, suspected or confirmed prostatitis, known ileal loops, or any of the following clinically significant laboratory abnormalities: absolute neutrophil count (ANC) <500 cells/µL, platelet count <40,000 cells/µL, serum alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin >5x the age-specific upper limit of normal (ULN), acute or chronic renal insufficiency with a baseline creatinine clearance <60 mL per minute or requires dialysis therapy for any reason
* Have a history of uncontrolled epilepsy defined as at least 1 seizure within the 6 months before randomization

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2010-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (38):
- United States (11):
  - Little Rock, Arkansas
  - Oakland, California
  - Orange, California
  - San Diego, California
  - Washington D.C., District of Columbia
  - New Brunswick, New Jersey
  - Albany, New York
  - The Bronx, New York
  - Cleveland, Ohio
  - Toledo, Ohio
  - Pittsburgh, Pennsylvania
- Argentina (4):
  - Buenos Aires
  - Córdoba
  - Loma Hermosa
  - Santa Fe
- Brazil (4):
  - Belo Horizonte
  - Caxias do Sul
  - Passo Fundo
  - São Paulo
- Chile (2):
  - Santiago
  - Valdivia X Región
- Colombia (4):
  - Bogotá
  - Cali
  - Floridablanca
  - Medellín
- Czechia (2):
  - Hradec Králové
  - Prague
- Riga, Latvia
- Lithuania (2):
  - Kaunas
  - Vilnius
- Mexico (3):
  - Guadajalara
  - Monterrey
  - Zapopan
- Zona, Panama
- Poland (2):
  - Lublin
  - Szczecin
- Ukraine (2):
  - Kharkiv
  - Poltava

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=3412&filename=CR100747_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Doripenem: Doripenem 20 mg/kg per dose (up to 500 mg/dose) was administered every 8 hours as 60-minutes IV (at least 3 days of IV doripenem only or IV doripenem followed by oral amoxicillin/clavulanate potassium or ciprofloxacin). Total duration of treatment 10 to 14 days.
- Cefepime: Cefepime 50 mg/kg per dose (up to 2 g/dose) was administered every 8 hours as 30-minutes IV (at least 3 days of IV cefepime only or IV cefepime followed by oral amoxicillin/clavulanate potassium or ciprofloxacin). Total duration of treatment 10 to 14 days.
Period: Overall Study
Arm/Group | Doripenem | Cefepime
Started | 31 | 10
Completed | 30 | 10
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doripenem | Cefepime | Total
Number analyzed (Participants) | 31 | 10 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31 | 10 | 41
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.7 (5.15) | 4.3 (4.16) | 4.6 (4.88)
Age, Customized [Number; unit: participants]
  3 months to <2 years | 12 | 4 | 16
  2 to <6 years | 8 | 2 | 10
  6 to <12 years | 7 | 3 | 10
  12 to <18 years | 4 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 5 | 31
  Male | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Clinical Cure Rate at Test Of Cure (TOC) Visit
Description: The participants were classified as cure if they had resolution or clinical improvement in signs and symptoms of complicated urinary tract infection; had no fever; no additional antimicrobial therapy was required for the treatment of the infection; and a clinical response assessment of improvement at End of IV visit.
Time Frame: TOC (7 to 14 days after the last dose of study medication therapy)
Population: Clinical Intent-to-Treat (CITT): All randomized participants who met the minimal disease definition of complicated urinary tract infection regardless if a baseline pathogen was isolated from the pretreatment urine culture.
Measure: Number; unit: Participants
Arm/Group | Doripenem | Cefepime
Number analyzed (Participants) | 30 | 10
Participants | 20 | 5

2. Secondary Outcome: The Number of Participants With Clinical Improvement Rate at End of IV (EIV) Visit
Description: The participants were considered as clinical improved if they had clinical improvement in signs and symptoms from baseline; no fever for at least the 24 hours before discontinuing the IV study drug; and not received nonstudy antibiotics for the treatment of urinary tract infection after IV study drug therapy had begun.
Time Frame: EIV (within 24 hours after completion of the last dose of IV study medication therapy)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Doripenem | Cefepime
Number analyzed (Participants) | 30 | 10
Participants | 28 | 10

3. Secondary Outcome: The Number of Participants With Clinical Cure Rate at Late Follow-Up (LFU) Visit
Description: The participants were classified as clinical cure if all pretreatment signs and symptoms of complicated urinary tract infection showed no evidence of recurrence after test of cure.
Time Frame: LFU (28 to 42 days after the last dose of study medication therapy)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Doripenem | Cefepime
Number analyzed (Participants) | 30 | 10
Participants | 18 | 5

4. Secondary Outcome: The Number of Participants With Favorable Per-participant Microbiological Response
Description: Favorable per-participant microbiological response rate was evaluated at the at End of IV (EIV) visit, Test Of Cure (TOC) visit, and Late Follow-Up (LFU) visit. The favorable per-participant microbiological response was considered when all baseline pathogens were eradicated (absence) or presumed eradicated (absence of material to culture in a participant who has a positive clinical response to treatment).
Time Frame: EIV (within 24 hours after completion of the last dose of IV study medication therapy), TOC (7 to 14 days after the last dose of study medication therapy), and LFU (28 to 42 days after the last dose of study medication therapy)
Population: Microbiological intent-to-treat - Participants of all CITT with at least 1 baseline bacterial pathogen isolated from the pretreatment urine culture, susceptible to both doripenem and cefepime. 6 and 2 participants from doripenem and cefepime, respectively had no susceptible urine pathogens at baseline and were excluded from this set.
Measure: Number; unit: Participants
Arm/Group | Doripenem | Cefepime
Number analyzed (Participants) | 24 | 8
Participants
  EIV visit | 24 | 8
  TOC visit | 19 | 4
  LFU visit | 16 | 4

5. Secondary Outcome: Number of Participants With Favorable Per-pathogen Microbiological Outcome Rate at End of IV (EIV) Visit
Description: The favorable per-pathogen microbiological outcome was considered when all baseline pathogens were eradicated (absence) or presumed eradicated (absence of material to culture in a participant who has a positive clinical response to treatment).A total of 4 pathogens in the doripenem group and 2 pathogens in the cefepime group were isolated at baseline from urine culture and were susceptible to the study drug received (see listed in the table below; the numbers in parenthesis next to each pathogen represent the number of participants with the pathogen isolated at baseline in the doripenem and cefepime treatment groups, respectively).
Time Frame: EIV (within 24 hours after completion of the last dose of IV study medication therapy)
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Doripenem | Cefepime
Number analyzed (Participants) | 24 | 8
Participants
  Staphylococcus aureus (3, 0) | 3 | NA — There were no participants with Stapylococcus aureus isolated at baseline.
  Escherichia coli (22, 7) | 22 | 7
  Klebsiella oxytoca (1, 0) | 1 | NA — There were no participants with Klebsiella oxytoca isolated at baseline.
  Klebsiella pneumoniae (1, 1) | 1 | 1

6. Secondary Outcome: Number of Participants With Favorable Per-pathogen Microbiological Outcome Rate at Test Of Cure (TOC) Visit
Description: The favorable per-pathogen microbiological outcome was considered when all baseline pathogens were eradicated (absence) or presumed eradicated (absence of material to culture in a participant who has a positive clinical response to treatment). A total of 4 pathogens in the doripenem group and 2 pathogens in the cefepime group were isolated at baseline from urine culture and were susceptible to the study drug received (see listed in the table below; the numbers in parenthesis next to each pathogen represent the number of participants with the pathogen isolated at baseline in the doripenem and cefepime treatment groups, respectively).
Time Frame: TOC (7 to 14 days after the last dose of study medication therapy)
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Doripenem | Cefepime
Number analyzed (Participants) | 24 | 8
Participants
  Staphylococcus aureus (3, 0) | 3 | NA — There were no participants with Stapylococcus aureus isolated at baseline.
  Escherichia coli (22, 7) | 17 | 4
  Klebsiella oxytoca (1, 0) | 1 | NA — There were no participants with Klebsiella oxytoca isolated at baseline
  Klebsiella pneumoniae (1, 1) | 1 | 0

7. Secondary Outcome: Number of Participants With Sustained Favorable Per-pathogen Microbiological Outcome Rate at Late Follow-Up (LFU) Visit
Description: The sustained favorable per-pathogen microbiological outcome was considered when all baseline pathogens were eradicated (absence) or presumed eradicated (absence of material to culture in a participant who has a positive clinical response to treatment). A total of 4 pathogens in the doripenem group and 2 pathogens in the cefepime group were isolated at baseline from urine culture and were susceptible to the study drug received (see listed in the table below; the numbers in parenthesis next to each pathogen represent the number of participants with the pathogen isolated at baseline in the doripenem and cefepime treatment groups, respectively).
Time Frame: LFU (28 to 42 days after the last dose of study medication therapy)
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Doripenem | Cefepime
Number analyzed (Participants) | 24 | 8
Participants
  Staphylococcus aureus (3, 0) | 2 | NA — There were no participants with Stapylococcus aureus isolated at baseline.
  Escherichia coli (22, 7) | 14 | 4
  Klebsiella oxytoca (1, 0) | 1 | NA — There were no participants with Klebsiella oxytoca isolated at baseline.
  Klebsiella pneumoniae (1, 1) | 1 | 0

ADVERSE EVENTS:
Time Frame: Approximately 8 weeks
Arm/Group | Doripenem | Cefepime
Serious Adverse Events (participants affected / at risk) | 1/30 | 3/10
Other Adverse Events (participants affected / at risk) | 11/30 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Doripenem (N=30) | Cefepime (N=10)
Pyuria (Renal and urinary disorders) | 1 | 0
Pseudomembranous Colitis (Infections and infestations) | 0 | 1
Pyelonephritis Acute (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Doripenem (N=30) | Cefepime (N=10)
Vomiting (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Pyrexia (General disorders) | 3 | 1
Infusion Site Pain (General disorders) | 0 | 1
Vessel Puncture Site Pain (General disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 0
Bacteriuria (Infections and infestations) | 0 | 1
Candidiasis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 1
Hypochromic Anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutrophilia (Blood and lymphatic system disorders) | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1
Congenital Thrombocyte Disorder (Congenital, familial and genetic disorders) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Basophil Count Increased (Investigations) | 0 | 1
Urine Leukocyte Esterase (Investigations) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Crystalluria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Leukocyturia (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This study was terminated early due to business reasons and not related to safety concerns or issues. As such, the limited enrollment precludes a meaningful conclusion about the efficacy and safety of doripenem compared with cefepime.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days